CLINICAL TRIAL: NCT01753102
Title: EFFICACY AND SAFETY OF SPIL'S ESTRADIOL VAGINAL TABLET, 10 MCG ESTRADIOL IN SUBJECTS WITH VULVAR AND VAGINAL ATROPHY: A RANDOMIZED, OBSERVER BLIND, PARALLEL GROUPS, ACTIVE AND PLACEBO CONTROLLED, CLINICAL ENDPOINT BIOEQUIVALENCE STUDY
Brief Title: Efficacy and Safety Of Spil's Estradiol Vaginal Tablet
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLR_10_19; CTRI/2012/09/002983 (Other: DCGI)
Record Dates: First submitted 2012-12-15; First posted 2012-12-20 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Vulvar Atrophy; Vaginal Atrophy
Keywords: Estradiol; Vulvar atrophy; vaginal atrophy
MeSH Terms: interventions — Estradiol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Estradiol (Experimental): Intravaginal self-administration of study medication once daily for 14 days.
  Interventions: Drug: Estradiol
- Reference: Estradiol (Active Comparator): Intravaginal self-administration of study medication once daily for 14 days.
  Interventions: Drug: Estradiol
- Placebo (Placebo Comparator): Intravaginal self-administration of study medication once daily for 14 days.
  Interventions: Drug: Estradiol

INTERVENTIONS:
Drug: Estradiol — one tablet will be inserted daily for 14 days
  Other Names: Vagifem

SUMMARY:
Estradiol vaginal tablet is a tablet which hydrates upon contact with moisture, releasing 17ß-estradiol.

The estradiol in estradiol vaginal tablet is chemically and biologically identical to the endogenous human estradiol and is therefore classified as a human estrogen.

The purpose of this study is to demonstrate clinical endpoint bioequivalence of SPIL's Estradiol vaginal tablet, 10mcg estradiol to the reference listed drug (Vagifem®)which is approved and marketed in the US.

DETAILED DESCRIPTION:
Estradiol vaginal tablet is indicated for use in the treatment of symptoms of atrophic vaginitis due to estrogen deficiency.

This is a randomized, observer blind, parallel groups, active and placebo controlled study to test the clinical endpoint bioequivalence of test product (Estradiol vaginal tablet, 10mcg of Sun Pharmaceutical Industries Ltd. India) relative to reference (Vagifem®, Estradiol vaginal tablet, 10mcg estradiol of Novo Nordisk) in treatment of vulvar and vaginal atrophy.

The patients will be administered with one tablet intravaginally daily for 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal woman
* At least one subject-self-assessed moderate to severe symptom of vulvar and vaginal atrophy
* ≤ 5% superficial cells on vaginal smear cytology
* Vaginal pH > 5.0

Exclusion Criteria:

* Consumption of estrogen alone or estrogen/progestin containing drug products.
* Allergy to estradiol or related products
* History of breast cancer and significant risk factors for endometrial cancer
* Abnormal genital bleeding

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2012-11-06 (Actual); Primary Completion 2013-04-30 (Actual); Study Completion 2013-04-30 (Actual)

PRIMARY OUTCOMES:
Vaginal pH | 14 days

SECONDARY OUTCOMES:
Symptoms of vulvar and vaginal atrophy | 14 days
  Each subject will specify identified most bothersome symptoms vaginal dryness, vaginal and/or vulvar irritation/ itching, dysuria, vaginal pain associated with sexual activity, vaginal bleeding associated with sexual activity) and self-evaluate the symptom on a pre-defined scale

CONTACTS AND LOCATIONS:
Locations (1):
- Biniwale Clinic Pvt. Ltd,, Pune, Maharashtra, India